CLINICAL TRIAL: NCT06189040
Title: Assessment of the Immunogenicity and Safety of Marketed Vaccines for COVID-19 After Regular Schedule and Adapted Vaccine Schedules and Routes: BNT162b2, mRNA-1273 Vaccine and ChAdOx1-S [Recombinant]
Brief Title: Immunogenicity After COVID-19 Vaccines in Adapted Schedules
Acronym: IMCOVAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Pierre Van Damme, Head of the Centre for the Evaluation of Vaccination (CEV), Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IMCOVAS
Record Dates: First submitted 2023-12-20; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Coronavirus Disease 2019; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; ChAdOx1 nCoV-19

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded up to the venous blood draw used to assess the primary endpoint (day 112 for the long-interval treatment arm, day 56 for all other treatment arms). Afterwards, participants were unblinded because the registration of all administered COVID-19 vaccines was required by the Belgian government.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- BNT162b2 regular schedule (Active Comparator): day 0: intramuscular administration of BNT162b2 (30µg) day 28: intramuscular administration of BNT162b2 (30µg)
  Interventions: Drug: BNT162b2 30µg
- BNT162b2 + mRNA-1273 schedule (Experimental): day 0: intramuscular administration of BNT162b2 (30µg) day 28: intramuscular administration of mRNA-1273 (100µg)
  Interventions: Drug: BNT162b2 30µg; Drug: mRNA-1273 100µg
- BNT162b2 + ChAdOx1-S schedule (Experimental): day 0: intramuscular administration of BNT162b2 (30µg) day 28: intramuscular administration of ChAdOx1-S [recombinant] (not less than 2.5x10^8 infectious units)
  Interventions: Drug: BNT162b2 30µg; Drug: ChAdOx1-S [Recombinant]
- BNT162b2 low dose schedule (Experimental): day 0: intramuscular administration of BNT162b2 (20µg) day 28: intramuscular administration of BNT162b2 (20µg)
  Interventions: Drug: BNT162b2 20µg
- BNT162b2 long-interval schedule (Experimental): day 0: intramuscular administration of BNT162b2 (30µg) day 84: intramuscular administration of BNT162b2 (30µg)
  Interventions: Drug: BNT162b2 30µg
- BNT162b2 intradermal schedule (Experimental): day 0: intradermal administration of BNT162b2 (6µg) day 28: intradermal administration of BNT162b2 (6µg)
  Interventions: Drug: BNT162b2 6µg
- mRNA-1273 regular schedule (Active Comparator): day 0: intramuscular administration of mRNA-1273 (100µg) day 28: intramuscular administration of mRNA-1273 (100µg)
  Interventions: Drug: mRNA-1273 100µg
- mRNA-1273 low dose schedule (Experimental): day 0: intramuscular administration of mRNA-1273 (50µg) day 28: intramuscular administration of mRNA-1273 (50µg)
  Interventions: Drug: mRNA-1273 50µg

INTERVENTIONS:
Drug: BNT162b2 30µg — intramuscular administration of 30µg
  Arms: BNT162b2 + ChAdOx1-S schedule; BNT162b2 + mRNA-1273 schedule; BNT162b2 long-interval schedule; BNT162b2 regular schedule
Drug: BNT162b2 20µg — intramuscular administration of 20µg
  Arms: BNT162b2 low dose schedule
Drug: BNT162b2 6µg — intradermal administration of 6µg
  Arms: BNT162b2 intradermal schedule
Drug: mRNA-1273 100µg — intramuscular administration of 100µg
  Arms: BNT162b2 + mRNA-1273 schedule; mRNA-1273 regular schedule
Drug: mRNA-1273 50µg — intramuscular administration of 50µg
  Arms: mRNA-1273 low dose schedule
Drug: ChAdOx1-S [Recombinant] — intramuscular administration of not less than 2.5 x 10^8 infectious units
  Arms: BNT162b2 + ChAdOx1-S schedule

SUMMARY:
The goal of this clinical trial is to compare different Coronavirus Disease 2019 (COVID-19) vaccination schedules in healthy adults that have not yet been exposed to SARS-CoV-2, the virus causing COVID-19. The main questions it aims to answer are:

1. Is it possible to adapt COVID-19 vaccination schedules while maintaining an adequate humoral immune response?
2. Is it possible to adapt COVID-19 vaccination schedules while maintaining an acceptable safety profile?

Participants will be vaccinated twice with a COVID-19 vaccine (on day 0, and on day 28 or 84). After each vaccination, they will collect information about adverse events in a diary for 14 days. Information about the occurrence of events such as hospitalizations and infections with SARS-CoV-2 will be collected by the investigator for up to 364 days after the first vaccination. Blood samples will be taken on different timepoints and used to assess immunity against SARS-CoV-2.

Researchers will compare 8 vaccination schedules to see if the immune response and safety profile is similar. Each participant will receive 1 of the following 8 vaccine schedules:

* BNT162b2 (30µg) on day 0, followed by BNT162b2 (30µg) on day 28
* BNT162b2 (20µg) on day 0, followed by BNT162b2 (20µg) on day 28
* BNT162b2 (30µg) on day 0, followed by BNT162b2 (30µg) on day 84
* BNT162b2 (30µg) on day 0, followed by mRNA-1273 (100µg) on day 28
* BNT162b2 (30µg) on day 0, followed by ChAdOx1-S [recombinant] on day 28
* BNT162b2 (6µg, intradermal administration) on day 0, followed by BNT162b2 (6µg, intradermal administration) on day 28
* mRNA-1273 (100µg) on day 0, followed by mRNA-1273 (100µg) on day 28
* mRNA-1273 (50µg) on day 0, followed by mRNA-1273 (50µg) on day 28

ELIGIBILITY:
Inclusion Criteria:

1. Male, female, or X (non-binary gender) subjects, 18-55y inclusive on the day of signing of the ICF
2. Provision of signed and dated informed consent form
3. Available at all provided timepoints of the study and is not planning to move abroad for the whole duration of the study
4. In good general health as evidenced by medical history and/or physical examination or adults with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
5. Willing and able to comply with all study procedures
6. Participants born female must be either:

   * of childbearing potential and using effective contraception for at least 1 month prior to screening and agree to use such a method during study participation until 1 months following the last study dose administration.
   * of non-childbearing potential.

Exclusion Criteria:

1. Previous clinical or microbiological confirmed diagnosis of COVID-19.
2. Febrile illness within 72hours before first vaccination (this is a temporary exclusion criterion).
3. Unstable, severe, progressive disease in the past 3 months.
4. History of malignancy during the past 5 years.
5. History of severe adverse reaction associated and/or anaphylaxis with a vaccine.
6. Known allergic reactions of any severity to polyethylene glycol [PEG] or to polysorbate (due to potential cross-reactive hypersensitivity with the vaccine ingredient PEG).
7. Primary or secondary immunodeficiency disorders (e.g. immunosuppressive disease or therapy, human immunodeficiency virus (HIV) infection…).
8. Chronic administration (defined as more than 14 days in total) of immunosuppressant or other immune-modifying drugs during the period starting 6 months prior to the first vaccine dose. For corticosteroids, this will mean prednisone 20 mg/day, or equivalent. Inhaled, nasal, opthalmic and topical steroids are allowed.
9. Pregnancy or lactation.
10. History of drug or alcohol abuse.
11. Anything in the opinion of the investigator that would prevent volunteers from completing the study or put the volunteer at risk, including relevant psychiatric diagnosis.
12. Previous vaccination or planned to accept other vaccination during this study with any coronavirus vaccine outside this study.
13. Previous vaccination or planned to accept other vaccination during this study with any coronavirus vaccine outside this study, with the exception of a third COVID-19 vaccine during fall/winter '21-'22.
14. Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
15. Participation in another clinical trial with an IMP or a new medical device within 28 days prior to study entry and/or during study participation.
16. Participant is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as first degree family members and household members of the employees or the investigator, or an employee of the sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 580 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Geometric mean titre of antibodies binding to the Receptor Binding Domain of SARS-CoV-2 S protein of the ancestral D614 SARS-CoV-2 virus strain | 28 days after the administration of the second study vaccine

SECONDARY OUTCOMES:
Occurrence of solicited adverse events | within 5 days after the administration of each study vaccine
Occurrence of unsolicited adverse events | within 14 days after the administration of each study vaccine
Occurrence of medically attended adverse events, adverse of special interest and serious adverse events | through study completion (up to 1 year after the first study vaccination)
Occurrence of absenteeism | within 5 days after the administration of each study vaccine
Geometric mean titre of antibodies binding to the Receptor Binding Domain of SARS-CoV-2 S protein of the ancestral D614 SARS-CoV-2 virus strain | 28 days after the administration of the third COVID-19 vaccine
Geometric mean titre of neutralizing antibodies to the ancestral D614 SARS-CoV-2 virus strain and variants of concern | 28 days after the administration of the second study vaccin
Geometric mean titre of neutralizing antibodies to the ancestral D614 SARS-CoV-2 virus strain and variants of concern | 28 days after the administration of the third COVID-19 vaccine

OTHER OUTCOMES:
PCR-confirmed SARS-CoV-2 infection with COVID-19 symptoms (any severity) | through study completion (up to 1 year after the first study vaccination)
PCR-confirmed SARS-CoV-2 infection with severe COVID-19 (hospitalization, death) | through study completion (up to 1 year after the first study vaccination)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Steenackers, MD, Principal Investigator — Centre for the Evaluation of Vaccination; Nikita Hanning, MD, Principal Investigator — Centre for the Evaluation of Vaccination
Locations (4):
- Belgium (4):
  - Centre for the Evaluation of Vaccination (CEV), Edegem, Antwerp
  - Centre for Vaccinology (CEVAC), Ghent, East Flanders
  - Institute of Tropical Medicine (ITM), Antwerp
  - Hôpital Erasme, Brussels

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analyzed during the current study are available from the central contact person on reasonable request, following material transfer agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Datasets will become available - upon request - after publication of the main results in a peer-reviewed scientific journal.
Access Criteria: The datasets used and analyzed during the current study are available from the central contact person on reasonable request, following material transfer agreements.

REFERENCES:
- [Derived] Steenackers K, Hanning N, Bruckers L, Desombere I, Marchant A, Arien KK, Georges D, Soentjens P, D'Onofrio V, Hites M, Berens-Riha N, De Coster I, Damme PV. Humoral immune response against SARS-CoV-2 after adapted COVID-19 vaccine schedules in healthy adults: The IMCOVAS randomized clinical trial. Vaccine. 2024 Nov 14;42(25):126117. doi: 10.1016/j.vaccine.2024.07.018. Epub 2024 Jul 16. PMID 39019657